CLINICAL TRIAL: NCT03758742
Title: Effect of Whole Fruit on Glycemic Control in Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Courtney M Peterson, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300001719; P30DK079626 (NIH)
Record Dates: First submitted 2018-11-16; First posted 2018-11-29 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; whole fruit; diabetes remission; glycemic control; liver fat; intrahepatic lipid; controlled feeding trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fatty Liver

STUDY DESIGN:
Masking Description: Lab values and week 0, 4, and 12 endpoints are assessed blinded by individuals not affiliated with the protocol. Also, data cleaning will be performed while being blinded to the timepoint.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-Fruit Diet (Experimental): Whole fruit-rich diet (~50% of calories from whole fruit)
  Interventions: Behavioral: High-Fruit Diet

INTERVENTIONS:
Behavioral: High-Fruit Diet — In this supervised controlled feeding study, participants will consume a diet rich in whole fruit. During the Ramp-Up Phase (Weeks 1-4), participants will gradually increase the amount of whole fruit they consume, eventually reaching 50% of calories from whole fruit. In the Main Phase (Weeks 5-12), participants will consume a whole fruit-rich, eucaloric diet that provides 50% of calories in the form of whole fruit. The non-fruit portion of the diet will be styled as a Mediterranean Diet. Participants will be required to approximately keep their weight stable throughout the intervention.

SUMMARY:
Diabetes costs the U.S. healthcare system more than any other disease, and nearly half of Americans will develop either diabetes or prediabetes in their lifetime. It is therefore critical to find new strategies to treat or reverse diabetes.

One such approach is adopting a healthy diet, which can dramatically improve blood sugar levels in adults with type 2 diabetes and even induce diabetes remission. Despite this, not much is known about which food groups are most effective at improving blood sugar levels in patients with diabetes.

Interestingly, of the various food groups, epidemiologic data suggests that whole fruit may be one of the most efficacious at both preventing type 2 diabetes and improving blood sugar in patients with type 2 diabetes. However, few clinical trials have investigated the effects of whole fruit on blood sugar control. This study will therefore be the first to determine the effects of increasing whole fruit as a food group in type 2 diabetes patients. This supervised controlled feeding trial will test whether consuming a diet rich in whole fruit for 12 weeks can improve glycemic control and cardiometabolic health in weight-stable adults with type 2 diabetes. The primary endpoint is glycemic control. Since changes in medication doses can skew the interpretation of glycemic outcomes, glycemic control will be assessed hierarchically (in descending order of importance) using (a) attainment of nondiabetic glycemia without medications (as a proxy for diabetes remission), (b) medication effect scores, (c) mean glucose during an oral glucose tolerance test, and (d) 24-hour mean glucose from continuous glucose monitoring. As secondary aims, this study will also test whether consuming a large amount of fructose in whole food form affects liver fat, pancreatic fat, and cardiovascular disease risk factors.

ELIGIBILITY:
Inclusion Criteria:

* 20-70 years old
* BMI ≤45.0 kg/m^2
* First diagnosed with type 2 diabetes within the past 6 years
* HbA1c between 6.0-9.5%%

Exclusion Criteria:

* On insulin
* Diagnosis of diabetes before age 18
* Estimated glomerular filtration rate < 45 ml/min per 1.732 m^2
* Heart attack in the past 6 months or severe or unstable heart failure
* On weight loss medication
* Change in the dosage of a chronic medication that may affect study endpoints within the past 3 months
* Clinically significant laboratory abnormality (e.g. abnormal hemoglobin levels)
* Significant gastrointestinal disease, major gastrointestinal surgery, or gallstones
* Significant cardiovascular, renal, cardiac, liver, lung, adrenal, or nervous system disease that might compromise safety or data validity
* Evidence of cancer (other than non-melanoma skin cancer) within the last 5 years
* Lost or gained more than 5 kg of weight in the past 6 months
* Pregnant, planning to become pregnant in the next 12 months, or breastfeeding
* Major psychiatric condition that would affect the ability to participate in the study
* Not able to eat the provided study meals
* Behavioral factors or circumstances that may impede adhering to the dietary intervention
* Not able to do the MRI/MRS abdominal scan, such as due to claustrophobia, implanted metal objects, or a body girth of 60 cm or greater

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney M. Peterson, Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Department of Nutrition Sciences, University of Alabamam at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Cobelli C, Dalla Man C, Toffolo G, Basu R, Vella A, Rizza R. The oral minimal model method. Diabetes. 2014 Apr;63(4):1203-13. doi: 10.2337/db13-1198. PMID 24651807
- [Derived] Hanick CJ, Berg KJ, Garvey WT, Goss AM, Steger FL, Richman JS, Peterson CM. Study protocol, menu design, and rationale for a study testing the effects of a whole fruit-rich diet on glycemic control, liver fat, pancreatic fat, and cardiovascular health in adults with type 2 diabetes. Nutr Res. 2025 Mar;135:82-100. doi: 10.1016/j.nutres.2025.01.008. Epub 2025 Jan 27. PMID 39978247

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-Fruit Diet
Started | 34
Completed | 12
Not Completed | 22

BASELINE CHARACTERISTICS:
Population: Results were analyzed only per-protocol, as is the norm for controlled feeding trials. In our study, per-protocol was defined as (a) completing the study with >=80% adherence and (b) meeting the weight stability criterion. Twelve participants completed the study, and of these, ten also met the weight stability criterion.
Groups:
- High-Fruit Diet: Whole fruit-rich diet (~50% of calories from whole fruit)
  High-Fruit Diet: Participants will consume a diet rich in whole fruit. During Phase I (Weeks 1-4; supervised controlled feeding), participants will gradually increase the amount of whole fruit they consume, eventually reaching 50% of calories from whole fruit. In Phase II (Week 5-12; supervised controlled feeding), participants will consume a whole fruit-rich, eucaloric diet that provides 50% of calories in the form of whole fruit. The non-fruit portion of the diet will be styled as a Mediterranean Diet. Participants will be required to approximately keep their weight stable during Phases I and II. In the Follow-Up Phase (Months 4-12; free-living), participants will be instructed to continue consuming at least one-third of their diet as whole fruit and to make healthy food choices.
Arm/Group | High-Fruit Diet
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Diabetes Remission Rate
Description: Percentage of patients who can maintain non-diabetic levels 24-hour mean glucose without the aid of pharmacotherapy at week 12
Time Frame: Change from baseline to week 12
Population: Results were analyzed per-protocol in completers who met the specified weight stability criterion
Measure: Count of Participants; unit: Participants
Groups:
- Fruit-Rich Diet: In this supervised controlled feeding study, participants will consume a diet rich in whole fruit. During the Ramp-Up Phase (Weeks 1-4), participants will gradually increase the amount of whole fruit they consume, eventually reaching 50% of calories from whole fruit. In the Main Phase (Weeks 5-12), participants will consume a whole fruit-rich, eucaloric diet that provides 50% of calories in the form of whole fruit. The non-fruit portion of the diet will be styled as a Mediterranean Diet. Participants will be required to approximately keep their weight stable throughout the intervention.
Arm/Group | Fruit-Rich Diet
Number analyzed (Participants) | 10
Participants
  % Who Maintained Non-Diabetic Glycemia Without Pharmacotherapy | 3
  % Who Weaned Off All Antihyperglycemic Medications | 6
Statistical Analysis 1: Comparison: Fruit-Rich Diet; Test type: Superiority; p < 0.0001, Binomial Test

2. Primary Outcome: Medication Effect Score (MES)
Description: % (or percentage). This quantity estimates the percentage by which all anithyperglycemic medications taken by a patient would lower HbA1c levels (i.e., percent of glycated hemoglobin molecules). Higher values indicate a higher dose and/or potency of medications.
Time Frame: Change from baseline to Week 12
Population: Results were analyzed per-protocol in completers who met the specified weight stability criterion
Measure: Least Squares Mean (Standard Error); unit: % (see definition under "Description")
Arm/Group | Fruit-Rich Diet
Number analyzed (Participants) | 10
% (see definition under "Description") | -0.5 (0.5)

3. Primary Outcome: Mean Glucose During a 3-hour Oral Glucose Tolerance Test (OGTT)
Description: mg/dl
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints). Change from week 0 to 12 reported.
Population: We present the results both in all participants (n=10) and those who were on stable doses of medications (n=4). The former data is presented for completeness only.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | High-Fruit Diet
Number analyzed (Participants) | 10
mg/dl
  All n=10 participants, including those who changed their medication doses | 11 (9)
  n=4 participants without medication changes: number analyzed (Participants) | 4
  n=4 participants without medication changes | -20 (12)

4. Primary Outcome: Mean 24-hour Glucose Levels as Measured by Continuous Glucose Monitoring (CGM), Adjusted for Any Changes in Medication Doses Via the MES
Description: mg/dl
Time Frame: as for outcome 3
Population: Results were analyzed per-protocol in completers who met the specified weight stability criterion
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Arm/Group | Fruit-Rich Diet
Number analyzed (Participants) | 10
mg/dl
  Main Analysis | -12 (7)
  Post Hoc Analysis Excluding 1 Outlier with Very Low C-peptide Levels: number analyzed (Participants) | 9
  Post Hoc Analysis Excluding 1 Outlier with Very Low C-peptide Levels | -18 (6)

5. Secondary Outcome: Insulin Sensitivity
Description: Insulin sensitivity (dl/kg/min/μU/ml) during a 3-hour OGTT, as measured by the Oral C-Peptide Minimal Model.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Error); unit: dl/kg/min/μU/ml
Arm/Group | High-Fruit Diet
Number analyzed (Participants) | 10
dl/kg/min/μU/ml
  All n=10 participants, including those who changed their medication doses | 1.27 (0.99)
  n=4 participants without medication changes: number analyzed (Participants) | 4
  n=4 participants without medication changes | 3.03 (1.61)

6. Secondary Outcome: Dynamic Beta-Cell Responsivity
Description: Phi_dynamic during a 3-hour OGTT, as measured by the Oral C-Peptide Minimal Model (which is a set of 5 coupled differential equations; see reference under Citations). Phi_dynamic is a measure of beta-cell responsiveness during first-phase insulin secretion. It is a dimensionless index (arbitrary units), where higher values denote greater insulin secretion.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Error); unit: arbitrary units * 10^9
Arm/Group | High-Fruit Diet
Number analyzed (Participants) | 10
arbitrary units * 10^9
  All n=10 participants, including those who changed their medication doses | 135 (60)
  n=4 participants without medication changes: number analyzed (Participants) | 4
  n=4 participants without medication changes | 122 (133)

7. Secondary Outcome: Static Beta-Cell Responsivity
Description: Phi_static during a 3-hour OGTT, as measured by the Oral C-Peptide Minimal Model (which is a set of 5 coupled differential equations; see reference under Citations). Phi_static is a measure of beta-cell responsiveness during second-phase insulin secretion. The units of measure are min^-1, and higher values denote greater insulin secretion.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Error); unit: 10^9/min
Arm/Group | High-Fruit Diet
Number analyzed (Participants) | 10
10^9/min
  All n=10 participants, including those who changed their medication doses | -3.0 (4.0)
  n=4 participants without medication changes: number analyzed (Participants) | 4
  n=4 participants without medication changes | 0.9 (10.6)

8. Secondary Outcome: Mean Insulin During a 3-hour OGTT
Description: mU/l
Time Frame: as for outcome 3
Population: We present the results both in all participants (n=10) and those who were on stable doses of medications (n=4). The former data is presented for completeness
Measure: Mean (Standard Error); unit: mU/l
Arm/Group | High-Fruit Diet
Number analyzed (Participants) | 10
mU/l
  All n=10 participants, including those who changed their medication doses | -17.1 (4.7)
  n=4 participants without medication changes: number analyzed (Participants) | 4
  n=4 participants without medication changes | -38.1 (6.7)

9. Secondary Outcome: Mean C-peptide During a 3-hour OGTT
Description: ng/ml
Time Frame: as for outcome 3
Population: as for outcome 8
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | High-Fruit Diet
Number analyzed (Participants) | 10
ng/ml
  All n=10 participants, including those who changed their medication doses | -0.4 (0.4)
  n=4 participants without medication changes: number analyzed (Participants) | 4
  n=4 participants without medication changes | -1.7 (0.5)

10. Secondary Outcome: Mean Amplitude of Glycemic Excursions From CGM
Description: mg/dl
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)"
Reporting Status: Not Posted

11. Secondary Outcome: Fasting Glucose
Description: mg/dl
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

12. Secondary Outcome: HbA1c
Description: percentage
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

13. Secondary Outcome: Liver Fat (Intrahepatic Lipid)
Description: Percentage as measured using Magnetic Resonance Spectroscopy (MRS) and 3-point M-Dixon Magnetic Resonance Imaging (MRI)
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

14. Secondary Outcome: Pancreatic Fat
Description: Percentage as measured using MRS and 3-point M-Dixon MRI methods
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

15. Secondary Outcome: Systolic and Diastolic Blood Pressure
Description: mm Hg
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

16. Secondary Outcome: Heart Rate
Description: beats per minute
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

17. Secondary Outcome: Time-in-range Metrics From CGM
Description: Time during which glucose levels are between 70 and 300 mg/dl
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

18. Secondary Outcome: Lipids
Description: Fasting total cholesterol (mg/dl), LDL cholesterol (mg/dl), HDL cholesterol (mg/dl), and triglycerides (mg/dl)
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Body Weight
Description: kg
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints); assessed weekly
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Waist Circumference
Description: cm
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Visceral Fat
Description: Visceral fat as measured using MRI (kg)
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Subcutaneous Abdominal Fat
Description: Subcutaneous abdominal fat as measured using MRI (kg)
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Gut Microbiome Diversity
Description: Diversity metrics (i.e., alpha and beta diversity)
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Gut Microbiome Composition
Description: Taxonomic composition and abundances
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Preference and Sensitivity to Sweet Tastes
Description: As measured on a 0-100 mm visual analog scale (VAS), using a Sweetness Taste Test
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Diet Satisfaction
Description: As measured on a 0-100 mm visual analog scale (VAS)
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Habitual Fruit Consumption
Description: As estimated using a series of semi-quantitative food frequency questions from the Diet History Questionnaire
Time Frame: Change from baseline to Weeks 4 and 12 and follow-up Months 6, 9, and 12
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Food Cravings
Description: As measured on five-point scales by the Food Craving Inventory-II
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Fruit Liking Visual Analog Scales
Description: As measured by VAS on a 0-100 mm scale
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Food Attitudes and Behaviors
Description: As measured by a modified version of the National Cancer Institute (NCI) 2007 Food Attitudes and Behaviors Survey, which covers constructs including attitudes and beliefs, fruit and vegetable consumption, eating behaviors, and food preferences
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

31. Other Pre Specified Outcome: General Health Status
Description: Healthy days (along various dimensions) as measured by the Centers for Disease Control and Prevention's (CDC) Health-Related Qualify of Life questionnaire
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Depression
Description: As measured on a 0-27 point scale by the Patient Health Questionnaire-9
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Mood States
Description: As measured on a 5-point scale by the Profile of Mood States Short-Form
Time Frame: Changes from weeks 0 to 12 (primary timepoint) and weeks 0 to 4 and 4 to 12 (secondary timepoints)
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Intervention Satisfaction and Feedback
Description: As measured by qualitative exit interview
Time Frame: Week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected at baseline (~1 week) and during Weeks 1 through 12.
Description: Participants were queried about adverse events at each study visit.
Arm/Group | High-Fruit Diet
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 18/34
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High-Fruit Diet (N=34)
Hypoglycemia (Metabolism and nutrition disorders) | 18 — <70 mg/dl
Hyperglycemia (Metabolism and nutrition disorders) | 15 — >300 mg/dl
Mild Stomach Pain (Gastrointestinal disorders) | 4
Mild Tremor (Nervous system disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 3
Fatigue (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03758742/Prot_SAP_000.pdf